CLINICAL TRIAL: NCT05663346
Title: Evaluation of a Digital Educational Intervention Regarding Safe and Efficient Cannabis Use with Young Adults Diagnosed with Cancer: a Pilot Study
Brief Title: Cannabis and Cancer, an Online Training for Oncology Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022-2802
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cannabis Use; Cannabis Use, Unspecified; Nurse's Role; Oncology Pain; Symptoms and Signs
MeSH Terms: conditions — Cancer Pain; Signs and Symptoms | interventions — nabiximols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis & Cancer digital educational intervention (Experimental): This intervention includes different asynchronous pedagogical modalities that allow, among other things, to reactivate the participants' previous knowledge and promote their autonomy in their learning process. These modalities focus on various problems that oncology nurses may encounter about the use of cannabis in oncology (eg, how to tackle the subject, what are the correct times to approach the topic). To this end, various pedagogical modalities that encourage the active participation of nurses are integrated into the training (eg, interactive videos, and quizzes). Scientific articles and links to external resources (official public websites) are also included so that nurses can consult the content at their own pace. Different aspects related to the use of cannabis are addressed in the training (eg, beneficial effects, and potential side effects).
  Interventions: Other: Cannabis & Cancer digital educational intervention
- Standard information regarding cannabis use in oncology (Active Comparator): The comparator is composed of an email with basic reliable non-personalized information on cannabis use in oncology (official public websites and scientific articles).
  Interventions: Other: Standard information regarding cannabis use in oncology

INTERVENTIONS:
Other: Cannabis & Cancer digital educational intervention — The Cannabis & Cancer intervention is available on Moodle learning management system in French language. It aims to influence nurses' self-efficacy, attitudes, intentions, and knowledge regarding the safe and efficient use of cannabis by young adults diagnosed with cancer.
  Arms: Cannabis & Cancer digital educational intervention
Other: Standard information regarding cannabis use in oncology — Participants will be offered basic reliable non-personalized information on cannabis use in oncology (official public websites and scientific articles).
  Arms: Standard information regarding cannabis use in oncology

SUMMARY:
The purpose of this study is to evaluate the preliminary effects and impacts of a digital educational intervention to support nurses' professional practice regarding safe cannabis use by young adults (18-39 years) diagnosed with cancer.

DETAILED DESCRIPTION:
This online pilot randomized controlled trial with parallel groups is conducted in Quebec (Canada). Moodle learning management system will be used to train nurses working in oncology.

After accepting the conditions and consenting, participants will enroll in the study by providing an email address. Each participant will be validated through an email address check. After their enrolment, participants will receive a hyperlink via email to invite them to complete a baseline questionnaire.

After completing the baseline questionnaire, participants will be randomly assigned by a research assistant to the digital educational intervention (Cannabis & Cancer) or to a control group (official public websites and scientific articles).

Four weeks after the baseline questionnaire, participants will complete the online questionnaires again.

ELIGIBILITY:
Inclusion Criteria:

* Work in an oncology department (eg, radio-oncology, outpatient clinics)
* Work with people diagnosed with cancer, including young adults
* Understand, read, and write French

Exclusion Criteria:

* None

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy | 4 weeks
  The French version of the Continuing Professional Development Reaction (CPD-Reaction) questionnaire (Légaré et al., 2014) will be used. The CPD-Reaction is a 12-item theory-based self-report questionnaire designed to assess the impact of continuing professional development on different clinical practices and can be modified according to the behavior targeted by the continuing professional activity (ie, the Cannabis & Cancer intervention).
  It is scored using a seven-point Likert scale ranging from strongly disagree (1) to strongly agree (7). The total score can range from 3 to 21 for self-efficacy. Higher scores indicate higher levels of self-efficacy. The CPD Reaction has adequate test-retest reliability (ie, weighted kappa coefficient between 0.43-0.53 for self-efficacy). The questionnaire has good internal consistency (Cronbach's alpha = 0.84).

SECONDARY OUTCOMES:
Change in attitudes | 4 weeks
  The French version of the Continuing Professional Development Reaction (CPD-Reaction) questionnaire (Légaré et al., 2014) will be used. The CPD-Reaction is a 12-item theory-based self-report questionnaire designed to assess the impact of continuing professional development on different clinical practices and can be modified according to the behavior targeted by the continuing professional activity (ie, the Cannabis & Cancer intervention).
  It is scored using a seven-point Likert scale ranging from strongly disagree (1) to strongly agree (7). The total score can range from 2 to 14 for attitudes. Higher scores indicate more favorable attitudes toward the behavior. The CPD Reaction has adequate test-retest reliability (ie, weighted kappa coefficient between 0.5-0.54 for attitudes). The questionnaire has good internal consistency (Cronbach's alpha = 0.89).
Change in intention | 4 weeks
  The French version of the Continuing Professional Development Reaction (CPD-Reaction) questionnaire (Légaré et al., 2014) will be used. The CPD-Reaction is a 12-item theory-based self-report questionnaire designed to assess the impact of continuing professional development on different clinical practices and can be modified according to the behavior targeted by the continuing professional activity (ie, the Cannabis & Cancer intervention).
  It is scored using a seven-point Likert scale ranging from strongly disagree (1) to strongly agree (7). The total score can range from 2 to 14 for intention. Higher scores indicate higher intentions to perform the behavior. The CPD Reaction has adequate test-retest reliability (ie, weighted kappa coefficient between 0.54-0.6 for intention). The questionnaire has good internal consistency (Cronbach's alpha = 0.79).
Change in knowledge | 4 weeks
  Nurses' knowledge will be assessed using a seven-point Likert scale (ie, 1=strongly disagree and 7=strongly agree) to be developed by the research team based on the educational content presented in the training.
Number of training modules completed by participants (objective engagement) | 4 weeks
  Objective data. This data will be collected automatically when users log into the learning management system.
Frequency of viewing modules/participants (objective engagement) | 4 weeks
  Objective data. This data will be collected automatically when users log into the learning management system.
Number of logins to the digital educational intervention/participant (objective engagement) | 4 weeks
  Objective data. This data will be collected automatically when users log into the learning management system.
Time required to complete all training modules (objective engagement) | 4 weeks
  Objective data. This data will be collected automatically when users log into the learning management system.
Subjective engagement with the digital educational intervention | 4 weeks
  Subjective engagement (self-reported) will be measured using the validated French version (Fontaine et al., 2020) of the User Engagement Scale - Short Form (UES-SF) (O'Brien et al., 2018). This 12-item instrument serves to measure four dimensions of engagement: 1) aesthetic appeal; 2) focused attention; 3) perceived usability, and 4) reward factor. Possible answers range from strongly disagree (+1) to strongly agree (+5). The possible total score ranges between 12 and 60. The score for each item will be interpreted and the scores for each dimension will be compared to indicate which are rated more highly than others. The French version shows acceptable internal consistency (ie, McDonald's omega coefficients ranging from 0.77-0.89).

CONTACTS AND LOCATIONS:
Overall Officials: Karine Bilodeau, PhD, Principal Investigator — Université de Montréal; José Côté, Principal Investigator — Université de Montréal; Billy Vinette, MSN, Principal Investigator — Univer
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vinette B, Cote J, Bilodeau K. Evaluation of a Digital Educational Intervention to Enhance Oncology Nurse Professional Practice to Support Safe Cannabis Use: A Pilot Study. J Contin Educ Health Prof. 2025 Dec 17. doi: 10.1097/CEH.0000000000000631. Online ahead of print. PMID 41427816